CLINICAL TRIAL: NCT00116259
Title: Aripiprazole in Children and Adolescents With Bipolar Disorder and ADHD: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Aripiprazole in Children and Adolescents With Bipolar Disorder and Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPPG03-325a; GPPG03-325a
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Bipolar Disorder; Attention Deficit Hyperactivity Disorder
Keywords: clinical trial; aripiprazole; Bipolar Disorder; Attention-Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Bipolar Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
There is a scarcity of clinical trials assessing the effects of medications in children with bipolar disorder. This study aims to assess the efficacy of Aripiprazole (a novel anti-psychotic drug) for the treatment of children and adolescents with bipolar disorder comorbid with ADHD. The study design is a 8-week randomized, double blind, parallel group trial. Patients were randomized to either aripiprazole or placebo.

The main hypotheses are:

1. Aripiprazole will significantly reduce maniac scores compared to placebo
2. Aripiprazole will significantly reduce ADHD scores compared to placebo

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic disorder that severely affects the normal development of children and adolescents. The disorder is associated with high rates of suicide tentative and high-risk behaviors like sexual promiscuity and drug abuse. Bipolar disorder in children is also associated with high rates of comorbidity, especially with Attention-Deficit Hyperactivity Disorder (ADHD). There is a scarcity of clinical trials assessing the effects of medications in children with BD. Moreover, the frequent presence of comorbid ADHD might determine lower response to treatment. Aripiprazole is a novel anti-psychotic drug. Its mechanism of action seems to be related to a stabilization of dopaminergic transmission, acting as a partial agonist especially in dopaminergic D2 receptors. It also has effects in 5-HT1a serotonergic receptors. Thus, it might have a promising effect in children and adolescents with comorbid BD and ADHD. A retrospective chart review, recently published, suggests the efficacy of this drug in children with BD. This study aims to assess the efficacy of Aripiprazole (a novel anti-psychotic drug) for the treatment of 50 children and adolescents (age range: 08 to 17 years-old) with Bipolar Disorder comorbid with ADHD. The study design is an 6-week randomized, double blind, parallel group trial. Patients were randomized to either aripiprazole or placebo. The hypotheses are: 1) Aripiprazole will significantly reduce maniac scores compared to placebo; 2)Aripiprazole will significantly reduce ADHD scores compared to placebo; 3) Aripiprazole will not be significantly associated to weight gain compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-17
* BD type I or II comorbid with ADHD
* Baseline score in the YMRS > or = 20

Exclusion Criteria:

* IQ < 70
* Pharmacologic treatment in the last month
* Pregnancy or absence of a contraceptive method in fertile girls
* Diagnoses: pervasive development disorder, schizophrenia, drug abuse or dependency
* Risk of suicide or homicide
* Clinical condition that might interfere in the study
* Known sensibility to aripiprazole

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Scores in the Young Mania Rating Scale (BD)
Scores in the SNAP-IV (ADHD)
Weight

SECONDARY OUTCOMES:
Scores in the CMRS-P
Scores in CGI
Scores in the CDRS
Scores in the Kutcher Adolescent Depression Scale
Scores of quality of life (YQOL-R)
Report of side events

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Rohde, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- ADHD outpatient program, Porto Alegre - Brazil, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Biederman J, McDonnell MA, Wozniak J, Spencer T, Aleardi M, Falzone R, Mick E. Aripiprazole in the treatment of pediatric bipolar disorder: a systematic chart review. CNS Spectr. 2005 Feb;10(2):141-8. doi: 10.1017/s1092852900019489. PMID 15685125
- [Derived] Tramontina S, Zeni CP, Ketzer CR, Pheula GF, Narvaez J, Rohde LA. Aripiprazole in children and adolescents with bipolar disorder comorbid with attention-deficit/hyperactivity disorder: a pilot randomized clinical trial. J Clin Psychiatry. 2009 Apr 21;70(5):756-64. doi: 10.4088/JCP.08m04726. PMID 19389329